CLINICAL TRIAL: NCT00978536
Title: A Monocenter, Cross-sectional Study to Compare Different Type of Cognitive Impairment in Multiple Sclerosis Patients and Cerebrospinal Fluid Biomarkers (Beta Amyloid, Total Tau Protein and Tau-phosphorylated Protein).
Acronym: BioCogS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties of recruitment in a randomization arm
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 08/11-K
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Disseminated Sclerosis
Keywords: Multiple sclerosis; cognitive deterioration; biomarkers; cerebrospinal fluid; Alzheimer disease
MeSH Terms: conditions — Multiple Sclerosis; Alzheimer Disease

ARMS (3):
- group 1 (Other): MS with cortical cognitive troubles
  Interventions: Other: Cognitive impairment of multiple sclerosis
- group 2 (Other): MS with subcortical cognitive troubles
  Interventions: Other: Cognitive impairment of multiple sclerosis
- group 3 (Other): MS in the early stage of the disease when cognitive troubles are absent or inconspicuous
  Interventions: Other: Cognitive impairment of multiple sclerosis

INTERVENTIONS:
Other: Cognitive impairment of multiple sclerosis — Patients will get a lumbar puncture in order to measure the biomarkers in the CSF, a neuropsychological exam, an evaluation of the hippocampal volume by MRI and a cerebral scintigraphy.

SUMMARY:
In multiple sclerosis (MS) sub cortical cognitive impairments are frequently reported. Nevertheless, cortical cognitive troubles, with hippocampic memory troubles have been described. Besides inflammatory damage, early cortical and degenerative damage are well known. In neurodegenerative diseases, three biomarkers of the cerebro spinal fluid (CSF), reflecting lesional mechanisms, are measured: the beta amyloid peptide, the tau total protein, and the phospho tau protein. Preliminary studies shown increased level of tau in MS. No study compare cognitive impairment and biomarkers of CSF.The aim of this study is to measure in the CSF of MS patients these three biomarkers (beta amyloid peptide, tau total and phosphotau) in order to establish correlations between a profile of biomarkers and a pattern of cognitive troubles, cortical or subcortical.The possibility to show, in MS patients with memory hippocampic troubles, a profile of biomarkers closed from the one encountered in AD, could argue in support of the degenerative hypothesis in MS and lead to discuss the interest of the use of AD treatment in MS.

ELIGIBILITY:
Inclusion Criteria:

* Groups 1 and 2 -patients MS - EDSS<7

Group 3- patients with first clinical inflammatory symptom

Exclusion Criteria:

* Pregnant or not taking contraceptive
* Contraindication for lumbar puncture
* Contraindication for NMR

Ages: 17 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The aim of this pilot study is to measure the level of total tau, phosphorylated tau and amyloid peptide in the CSF in order to establish correlations between a profile ofCSF biomarkers and a type of cognitive impairment, cortical or subcortical. | 15 months

SECONDARY OUTCOMES:
To compare each biomarker individually between the three groups. | 15 months
To define clinical and paraclinical characteristics of MS patients with cortical cognitive dysfunction by a clinical and neuropsychological evaluation, a morphological (cerebral MRI) and a functional exam (cerebral scintigraphy). | 15 Months

CONTACTS AND LOCATIONS:
Overall Officials: Claire Boutoleau-Bretonniere, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France